CLINICAL TRIAL: NCT06847529
Title: Systemic Inflammatory Markers As a Prognostic Index for B-cell Neoplasm , Single Center Experience .
Brief Title: Systemic Inflammatory Markers in B-cell Neoplasm
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marline Wiliam Fayez Abdel-Shahid, Resident Doctor, Assiut University
Other Study IDs: markers In B-cell tumors
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: B-cell Neoplasm
Keywords: Systemic inflammatory markers as a prognostic index
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study was to evaluate the role of systemic inflammatory markers in predicting outcome for patients with B cell neoplasm

DETAILED DESCRIPTION:
In malignant tumors, Inflammation plays a crucial role in the development, invasion, and metastasis of malignant tumors. Cancer is often described as a wound that does not heal, highlighting the significance of inflammation in cancer progression. Many tumors are heavily infiltrated by immune cells, including macrophages, neutrophils, and lymphocytes. Therefore, markers related to inflammation and the host immune response are pertinent as biological indicators of B-cell neoplasm progression. Inflammation contributes significantly to the initiation and advancement of B-cell neoplasms by providing nutrients to tumor cells, promoting cell growth, and disrupting immune homeostasis. Various composite indices based on circulating inflammatory cells have been developed as straightforward measures to assess systemic inflammation. Elevated serum inflammatory markers reflect the body's response to malignant tumors. Pro-inflammatory cytokines and inflammatory cells within the tumor microenvironment have been shown to promote tumor growth, induce DNA damage, facilitate angiogenesis, suppress the immune system, and correlate with poor patient survival outcomes. Targeting cytokine receptors or other components in inflammatory pathways involved in metastasis may offer therapeutic potential for malignant tumors. Given the pivotal role of inflammation in cancer biology, identifying novel immune markers is essential for predicting the prognosis of patients with Diffuse Large B-Cell Lymphoma (DLBCL). patients

ELIGIBILITY:
Inclusion Criteria:

* Individuals newly diagnosed with B-cell neoplasms, including:
* Burkitt's lymphoma (BL)
* Chronic lymphocytic leukemia (CLL)
* Diffuse large B-cell lymphoma (DLBCL)
* Follicular lymphoma (FL)
* Hairy cell leukemia (HCL)
* Splenic B-cell lymphoma/leukemia with prominent nucleoli (SBLPN)
* High-grade B-cell lymphoma (HGBL)
* Lymphoplasmacytic lymphoma (LPL)/Waldenström macroglobulinemia
* Mantle cell lymphoma (MCL)
* Splenic marginal zone lymphoma (MZL)
* Monoclonal B-cell lymphocytosis (MBL)
* Multiple myeloma (plasma cell myeloma)
* Monoclonal gammopathy of undetermined significance (MGUS)
* Age 18 years or older.

Exclusion Criteria:

* Individuals previously diagnosed with B-cell neoplasms.
* Individuals younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on determining the main outcome variable, the estimated minimum required sample size is 74. The sample size was calculated using G*power software 3.1.9.4 , based on the following assumptions: Main outcome variable is the evaluation of role of systemic inflammatory markers in predicting outcome for patients with B cell neoplasm. Based on expert opinion we hypothesized to find medium effect size 0.3
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-22 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Determination of Optimal Cut-off Values for Systemic Inflammatory Indices in B-cell Neoplasms Using Laboratory Blood Tests | Baseline
  This outcome measure aims to establish the optimal cut-off values for systemic inflammatory indices-including Neutrophil-to-Lymphocyte Ratio (NLR), Platelet-to-Lymphocyte Ratio (PLR), and Lymphocyte-to-Monocyte Ratio (LMR)-using routine laboratory blood tests. The blood tests will include serum lactate dehydrogenase (LDH), globulin, albumin, C-reactive protein (CRP), platelet count, neutrophil count, lymphocyte count, and monocyte count. Receiver Operating Characteristic (ROC) curve analysis will be employed to determine the optimal cut-off values for each inflammatory marker.

SECONDARY OUTCOMES:
Prognostic Value of Baseline Systemic Inflammatory Markers on Overall Survival in B-cell Neoplasm Patients | From baseline up to 8 months
  This outcome measure evaluates the association between baseline systemic inflammatory markers and overall survival in patients with B-cell neoplasms. The markers to be assessed include serum levels of LDH, globulin, albumin, CRP, and blood cell counts (neutrophils, lymphocytes, monocytes). Additionally, calculated indices such as NLR, PLR, LMR, CRP-to-Albumin Ratio (CAR), Albumin-to-Globulin Ratio (AGR), Systemic Immune-Inflammation Index (SII), and Systemic Inflammation Response Index (SIRI) will be determined. Patient follow-up will be conducted for 6 to 8 months or until the completion of the chemotherapeutic regimen or death.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Din Abdel Moneim El-Sayed, Doctor, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elinav E, Nowarski R, Thaiss CA, Hu B, Jin C, Flavell RA. Inflammation-induced cancer: crosstalk between tumours, immune cells and microorganisms. Nat Rev Cancer. 2013 Nov;13(11):759-71. doi: 10.1038/nrc3611. PMID 24154716
- [Background] Liu FT, Jia L, Wang P, Farren T, Li H, Hao X, Agrawal SG. CD126 and Targeted Therapy with Tocilizumab in Chronic Lymphocytic Leukemia. Clin Cancer Res. 2016 May 15;22(10):2462-9. doi: 10.1158/1078-0432.CCR-15-1139. Epub 2015 Dec 28. PMID 26712690
- [Background] Drutskaya MS, Nosenko MA, Atretkhany KS, Efimov GA, Nedospasov SA. [Interleukin-6 From molecular mechanisms of signal transduction to physiological properties and therapeutic targeting]. Mol Biol (Mosk). 2015 Nov-Dec;49(6):937-43. doi: 10.7868/S0026898415060063. Russian. PMID 26710772
- [Background] Goumas FA, Holmer R, Egberts JH, Gontarewicz A, Heneweer C, Geisen U, Hauser C, Mende MM, Legler K, Rocken C, Becker T, Waetzig GH, Rose-John S, Kalthoff H. Inhibition of IL-6 signaling significantly reduces primary tumor growth and recurrencies in orthotopic xenograft models of pancreatic cancer. Int J Cancer. 2015 Sep 1;137(5):1035-46. doi: 10.1002/ijc.29445. Epub 2015 Jan 29. PMID 25604508
- [Background] Kurzrock R, Voorhees PM, Casper C, Furman RR, Fayad L, Lonial S, Borghaei H, Jagannath S, Sokol L, Usmani SZ, van de Velde H, Qin X, Puchalski TA, Hall B, Reddy M, Qi M, van Rhee F. A phase I, open-label study of siltuximab, an anti-IL-6 monoclonal antibody, in patients with B-cell non-Hodgkin lymphoma, multiple myeloma, or Castleman disease. Clin Cancer Res. 2013 Jul 1;19(13):3659-70. doi: 10.1158/1078-0432.CCR-12-3349. Epub 2013 May 9. PMID 23659971
- [Background] Beguelin W, Sawh S, Chambwe N, Chan FC, Jiang Y, Choo JW, Scott DW, Chalmers A, Geng H, Tsikitas L, Tam W, Bhagat G, Gascoyne RD, Shaknovich R. IL10 receptor is a novel therapeutic target in DLBCLs. Leukemia. 2015 Aug;29(8):1684-94. doi: 10.1038/leu.2015.57. Epub 2015 Mar 3. PMID 25733167
- [Background] Marri PR, Hodge LS, Maurer MJ, Ziesmer SC, Slager SL, Habermann TM, Link BK, Cerhan JR, Novak AJ, Ansell SM. Prognostic significance of pretreatment serum cytokines in classical Hodgkin lymphoma. Clin Cancer Res. 2013 Dec 15;19(24):6812-9. doi: 10.1158/1078-0432.CCR-13-1879. Epub 2013 Oct 18. PMID 24141626
- [Background] Zhang L, Yang J, Qian J, Li H, Romaguera JE, Kwak LW, Wang M, Yi Q. Role of the microenvironment in mantle cell lymphoma: IL-6 is an important survival factor for the tumor cells. Blood. 2012 Nov 1;120(18):3783-92. doi: 10.1182/blood-2012-04-424630. Epub 2012 Sep 11. PMID 22968454
- [Background] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Background] Diakos CI, Charles KA, McMillan DC, Clarke SJ. Cancer-related inflammation and treatment effectiveness. Lancet Oncol. 2014 Oct;15(11):e493-503. doi: 10.1016/S1470-2045(14)70263-3. PMID 25281468
- [Background] Carbone A, Tripodo C, Carlo-Stella C, Santoro A, Gloghini A. The role of inflammation in lymphoma. Adv Exp Med Biol. 2014;816:315-33. doi: 10.1007/978-3-0348-0837-8_12. PMID 24818728
- [Background] Hogfeldt T, Bahnassy AA, Kwiecinska A, Osterborg A, Tamm KP, Porwit A, Zekri AR, Lundahl J, Khaled HM, Mellstedt H, Moshfegh A. Patients with activated B-cell like diffuse large B-cell lymphoma in high and low infectious disease areas have different inflammatory gene signatures. Leuk Lymphoma. 2013 May;54(5):996-1003. doi: 10.3109/10428194.2012.738365. Epub 2012 Nov 8. PMID 23046110
- [Background] Rotaru I, Gaman GD, Stanescu C, Gaman AM. Evaluation of parameters with potential prognosis impact in patients with primary gastric diffuse large B-cell lymphoma (PG-DLBCL). Rom J Morphol Embryol. 2014;55(1):15-21. PMID 24715160
- [Background] Eiro N, Vizoso FJ. Inflammation and cancer. World J Gastrointest Surg. 2012 Mar 27;4(3):62-72. doi: 10.4240/wjgs.v4.i3.62. PMID 22530080